CLINICAL TRIAL: NCT01094691
Title: Polyomavirus Aggregates, Haufen, in Voided Urine Samples as Diagnostic Biomarkers of Intra Renal BK-virus Disease: a Prospective Proof-of-concept Study
Brief Title: Haufen Diagnostic Biomarkers of BK Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-1519
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Polyoma Virus Nephropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Allograft Biopsy (Experimental): Urine left over from clinic visits is analyzed for 'Haufen' by negative staining electron microscopy as a marker of intra-renal polyomavirus nephropathy. Correlate Haufen, urine, and plasma data with the clinical presentation and with renal biopsy findings. Patients with PVN will be approached for study participation in which their routine samples will be monitored until urine is negative for 'Haufen', and a study protocol biopsy will be obtained for confirmation.
  Interventions: Procedure: Renal Allograft Biopsy

INTERVENTIONS:
Procedure: Renal Allograft Biopsy — A renal allograft biopsy will be performed when the urine is determined to be Haufen negative.

SUMMARY:
To prospectively test whether the detection of three-dimensional, cast-like polyomavirus aggregates, termed Haufen, in voided urine samples can serve as an accurate biomarker of intra-renal disease, i.e. polyoma-BK-virus nephropathy (PVN). We want to correlate the detection of 'Haufen' with histologic findings made in renal biopsies as well as signs of polyomavirus activation, i.e. viremia and viruria. The prospective study is designed to further validate our retrospective findings (manuscript in press, J Am Soc Nephrology) and more specifically to correlate 'Haufen' shedding with the histologically confirmed course of PVN.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Recipient of renal transplant
* Positive for polyoma virus
* Haufen cells present in urine
* Positive for polyoma virus nephropathy

Exclusion Criteria:

* anyone who does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Correlate Haufen, urine and plasma data with the clinical presentation and - in selected cases - with renal biopsy findings. | The biopsy will be performed when urine is determined to be Haufen negative

CONTACTS AND LOCATIONS:
Overall Officials: Volker Nickeleit, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-CH Dept of Pathology, Chapel Hill, North Carolina, United States